CLINICAL TRIAL: NCT00204880
Title: Aging and Cancer: The Effects of Comorbidities on Cancer and it's Treatment
Brief Title: Aging and Cancer Effects (ACE) Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0341
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypotheses:

1. Subjective self-reported data can be used to accurately reflect functioning across the 5 key domains.
2. Cancer and its various treatment modalities will exert detrimental effects on the 5 key domains in older adults with cancer.
3. Some aspect of baseline patient characteristic will be predictive of cancer-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to do memory testing
* Willing to participate in activities of daily living assessment
* Can use a cane or walker
* Willing to complete a balance performance assessment, if able.

Exclusion Criteria:

* Currently receiving treatment for cancer.
* Has a previous history of brain cancer
* Significant neurological disease other than AD that might affect cognitive function, such as stroke, Parkinson's disease, multiple sclerosis, or serious traumatic brain injury.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over the age of 55 newly diagnosed with lung, breast, colon or rectal cancer, and with an anticipated life expectancy of at least 2 years for breast cancer patients,1 year for patients with lung cancer, and 2 years for patients with colon or rectal cancer. There is no upper age limit for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2005-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Asthana, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States